CLINICAL TRIAL: NCT06651996
Title: Adherence and Feasibility of Remote Rehabilitation for Chronic Patellofemoral Joint Pain: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2023699
Record Dates: First submitted 2024-09-19; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: Patellofemoral Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- one session of face-to-face telerehabilitation tutorial (OST) (Sham Comparator): Participants were assigned to receive either one session of face-to-face telerehabilitation tutorial (OST) and complete an 8-week home digital health program consisting of sensor-guided exercise therapy and knee pain self-care education. The primary outcome was short-term adherence as assessed by the Exercise Adherence Rating Scale (EARS) after 6 weeks of face-to-face therapy. Secondary measures included pain intensity, quadriceps strength, Kujala patellofemoral score, fatigue severity scale, and qualitative interviews affecting adherence.
  Interventions: Device: one session of face-to-face telerehabilitation tutorial (OST)
- Three session of face-to-face telerehabilitation tutorials (TST) (Experimental): Participants were assigned to receive 3 in-person remote rehabilitation coaching (TST) sessions and complete an 8-week home digital health program consisting of sensor-guided exercise therapy and knee pain self-care education. The primary outcome was short-term adherence as assessed by the Exercise Adherence Rating Scale (EARS) after 6 weeks of face-to-face therapy. Secondary measures included pain intensity, quadriceps strength, Kujala patellofemoral score, fatigue severity scale, and qualitative interviews affecting adherence.
  Interventions: Device: Three session of face-to-face telerehabilitation tutorials (TST)
- Six session of face-to-face telerehabilitation tutorials (SST) (Experimental): Participants were assigned to receive 6 in-person remote rehabilitation coaching (SST) sessions and complete an 8-week home digital health program consisting of sensor-guided exercise therapy and knee pain self-care education. The primary outcome was short-term adherence as assessed by the Exercise Adherence Rating Scale (EARS) after 6 weeks of face-to-face therapy. Secondary measures included pain intensity, quadriceps strength, Kujala patellofemoral score, fatigue severity scale, and qualitative interviews affecting adherence.
  Interventions: Device: Six session of face-to-face telerehabilitation tutorials (SST)

INTERVENTIONS:
Device: one session of face-to-face telerehabilitation tutorial (OST) — The first group participated in a face-to-face tele-rehabilitation session in the hospital on the use of sensors and rehabilitation software before the home-rehabilitation session. Thereafter, the tele-rehabilitation program included muscle strengthening, flexibility stretching, and movement quality training every Tuesday, Thursday, and Saturday.
  Arms: one session of face-to-face telerehabilitation tutorial (OST)
Device: Three session of face-to-face telerehabilitation tutorials (TST) — The second group participated in three face-to-face tele-rehabilitation sessions in the hospital on the use of sensors and rehabilitation software before the home-rehabilitation session. Thereafter, the tele-rehabilitation program included muscle strengthening, flexibility stretching, and movement quality training every Tuesday, Thursday, and Saturday.
  Arms: Three session of face-to-face telerehabilitation tutorials (TST)
Device: Six session of face-to-face telerehabilitation tutorials (SST) — The third group participated in six face-to-face tele-rehabilitation sessions in the hospital on the use of sensors and rehabilitation software before the home-rehabilitation session. Thereafter, the tele-rehabilitation program included muscle strengthening, flexibility stretching, and movement quality training every Tuesday, Thursday, and Saturday.
  Arms: Six session of face-to-face telerehabilitation tutorials (SST)

SUMMARY:
This study is a prospective, single-center trial involving 66 patients diagnosed with patellofemoral pain. The study adhered to ethical guidelines and obtained informed consent from all participants. Participants were randomly assigned to receive face-to-face remote rehabilitation guidance either 1 time, 3 times, or 6 times. The primary outcome measure was exercise adherence assessed using the Exercise Rating Scale (EARS) after 6 weeks of rehabilitation. Secondary outcomes included knee pain severity, muscle strength, knee function, fatigue levels, and a qualitative research questionnaire. An isokinetic strength testing system was used to measure the open-chain strength of the quadriceps muscle.

DETAILED DESCRIPTION:
The inestigators conducted a forward-looking, single-center pilot study with a follow-up period of 8 weeks. The study recruited 66 patients diagnosed with patellofemoral pain (PFP) by a professional sports physician at the Department of Sports Medicine, Peking University Third Hospital, between January and September 2023. The study adhered to the principles of the Declaration of Helsinki and was approved by the Research Ethics Committee of Peking University Third Hospital. Although this is a pilot study, the inestigators strictly followed the CONSORT guidelines. All participants signed an informed consent form and completed home rehabilitation interventions.

Inclusion and Exclusion Criteria During the trial, an investigator not involved in the study used an electronically generated random sequence to assign patients to three groups. Two professional physical therapists (N.C and S.R) were responsible for assessing and supervising the accuracy of the project and were unaware of the grouping details.

Interventions After randomization, participants received a package containing two wearable motion sensors, a charger, resistance bands, and a manual. Additionally, the rehabilitation software provided lectures and Q&A sessions related to the condition, accessible via Android or iOS platforms. All data collected by the sensors were strictly encrypted to protect patient information and privacy. Each participant was assigned a therapist for home rehabilitation support, and a follow-up function via the software or telephone was used to remind patients who missed three remote rehabilitation sessions.

Before starting home rehabilitation, patients attended a briefing at the hospital. Participants were divided into three groups: Group 1 received 1 face-to-face remote rehabilitation tutorial (OST), Group 2 received 3 face-to-face remote rehabilitation tutorials (TST), and Group 3 received 6 face-to-face remote rehabilitation tutorials (SST). Each session lasted 40 minutes and was conducted three times a week (on Tuesday, Thursday, and Saturday). Following the briefing, patients performed home remote rehabilitation training on the same day, with each session lasting 40 minutes. The remote rehabilitation program included muscle strengthening, flexibility stretching, and movement quality training.

Primary Outcome The primary outcome was assessed by the Exercise Adherence Rating Scale (EARS) 6 weeks after completing the rehabilitation guidance. The scale consists of Part A, which directly assesses adherence (including 6 questions, each with 5 options, scoring from 0 to 4), and Part B, which assesses reasons affecting adherence (including 10 questions, each with 5 options, scoring from 0 to 4). Items with positive phrasing were reverse scored, so a higher overall adherence score indicates better exercise adherence.

Secondary Outcomes Secondary outcomes were collected at the hospital 8 weeks after the start of the study, including knee pain severity assessed by the Visual Analog Scale (VAS) (ranging from 0 "no pain" to 10 "worst pain"); isokinetic concentric and eccentric peak torque of the quadriceps muscle reflecting knee joint muscle strength; Kujala Patellofemoral Score (0 to 100 points, with higher scores indicating better knee function); and the Fatigue Severity Scale (FSS), which measures the severity of fatigue in patients with various conditions and its impact on activities and lifestyle (including 9 questions, each scored from 1 to 7, with higher scores indicating greater fatigue). Additionally, after completing the remote rehabilitation program, the inestigators conducted a qualitative research questionnaire to explore potential strategies to improve adherence.

ELIGIBILITY:
Inclusion Criteria:

* (1) Anterior knee pain or retro-patellar pain caused by at least two of the following activities: prolonged sitting with knee flexion, bilateral squatting, ascending and descending stairs, kneeling, running, and jumping;
* (2) presence of one of the following signs: patellar tenderness, friction pain, or twitching pain, positive single-leg squat test, or positive knee extension resistance test;
* (3) knee pain lasting more than 3 months;
* (4) knee pain score greater than 3 out of 10 on the VAS;
* (5) unilateral pain and symptoms.

Exclusion Criteria:

* (1) acute injury of the knee ligaments, joint capsule, bursa or meniscus;
* (2) knee extension or flexion contracture deformity, thus being unable to perform normal lower limb flexion and extension;
* (3) patellofemoral joint dislocation or subluxation;
* (4) any traumatic, inflammatory or infectious disease of the lower limbs;
* (5) a history of knee surgery;
* (6) a history of cardiovascular and cerebrovascular diseases, diabetes, tumors;
* (7) spinal cord or neurological injury.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-10-27 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure was the Exercise Adherence Rating Scale (EARS) at 6 weeks after the completion of the rehabilitation tutorial. | Six weeks after completion of face-to-face rehabilitation instruction
  The primary outcome measure was the Exercise Adherence Rating Scale (EARS) at 6 weeks after the completion of the rehabilitation tutorial. Section A directly evaluates the adherence (6 questions, 5 options per question represent 0-4 points), and Section B evaluates the reasons affecting the adherence (10 questions, 5 options per question represent 0-4 points. Positively phrased items were reversed scored so that a higher overall adherence score indicated better adherence to exercise)

SECONDARY OUTCOMES:
pain intensity | eight weeks after completion of face-to-face rehabilitation instruction
  Secondary outcome measures were collected at the hospital 8 weeks after the start of the study, including the severity of knee pain during daily living and squatting at 60 degrees (from 0 "no pain" to 10 "most severe") assessed on the visual analogue scale (VAS);
quadriceps strength | Eight weeks after the start of the trial
  Isokinetic quadriceps femoris concentric and eccentric peak torque reflect muscle strength around the knee joint.The open-chain muscle strength of the quadriceps muscle was tested with an isokinetic muscle strength testing system (Contrex MJ) in two modes: 60°/s centripetal contraction and 60°/s centrifugal contraction. The range of the test was from 90° to 20° of knee flexion. During the test, the subjects were asked to relax as much as possible before the test, with the trunk flexed at an angle of 120°, so that the test could be performed under the reduced influence of gravity. Each contraction mode was repeated 5 times, and the interval between adjacent contraction modes was 3 minutes to rest the thigh muscles.
Kujala scores | Eight weeks after the start of the trial
  Kujala patellofemoral score is used to evaluate the function of the knee joint (0-100, with higher scores indicating better knee function)
Fatigue severity scale | Eight weeks after the start of the trial
  Fatigue severity scale (FSS) is used to measure the fatigue degree of patients with various diseases and its impact on people's activities and lifestyle (9 questions in total, 7 points for each question, the higher the score, the greater the fatigue degree)
qualitative study questionnaire | Eight weeks after the start of the trial
  Furthermore, a qualitative study questionnaire was carried out post-completion of the tele-rehabilitation program to identify potential strategies for enhancing adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital Medicial Science Research Ethics Committee, Beijing, China

IPD SHARING:
Plan to Share IPD: No